CLINICAL TRIAL: NCT00203515
Title: A Prospective, Randomized, Controlled Study Comparing the DOVER Silver Foley Catheter to a Standard of Care Catheter and a Marketed Silver Coated Foley Catheter
Brief Title: Study Comparing the DOVER Silver Foley Catheter to a Standard of Care Catheter and a Marketed Silver Coated Foley Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tyco Healthcare Group (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 302.18
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2008-01

CONDITIONS: Urinary Tract Infections
Keywords: Urinary Catheterization
MeSH Terms: conditions — Urinary Tract Infections

INTERVENTIONS:
Device: Standard Latex Foley Catheter
Device: Silver Coated Latex Foley Catheter

SUMMARY:
The purpose of the study is to determine if the commercially available device called the DOVER™ Silver Foley catheter prevents infections of the urinary tract.

DETAILED DESCRIPTION:
Over 1 million catheter-associated urinary tract infections (CAUTIs) occur annually in U.S. healthcare facilities and account for approximately 40% of the nosocomial infections. This investigation is a multi-center, blinded, prospective, randomized, controlled, parallel comparison of the intervention catheter (Tyco Healthcare DOVER Silver Foley catheter) to a usual care catheter and another commercially available silver-coated catheter. 1000 subjects total will be randomized at the multiple study centers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* Subject is expected to be catheterized with a 14, 16 or 18 French Foley catheter for at least 72 hours.
* Subject or his/her legally authorized representative is able to grant informed consent to participate in this investigation.

Exclusion Criteria:

* Subjects who present with ongoing, active, symptomatic UTI.
* Subjects with a known or suspected allergy to silver or silver compounds causing delayed hypersensitivity reactions or contact dermatitis.
* Subjects with a known or suspected allergy to natural rubber latex or natural rubber latex compounds causing delayed hypersensitivity reactions or contact dermatitis.
* Subjects known to be pregnant.
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2005-01; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Catheter associated urinary tract infection (UTI)

SECONDARY OUTCOMES:
Catheter tolerance
Cost of care

CONTACTS AND LOCATIONS:
Overall Officials: Bethany A Quinn, Study Director — Tyco Healthcare Group/Kendall
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Background] Tambyah PA, Maki DG. The relationship between pyuria and infection in patients with indwelling urinary catheters: a prospective study of 761 patients. Arch Intern Med. 2000 Mar 13;160(5):673-7. doi: 10.1001/archinte.160.5.673. PMID 10724053